CLINICAL TRIAL: NCT05797298
Title: Plate-haptic Toric Intraocular Lens (IOL) Implantation for Management of Cataracts
Brief Title: Toric Intraocular Lens (IOL) Implantation for Management of Cataracts
Status: Recruiting | Type: Observational
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Other Study IDs: Toric IOL
Record Dates: First submitted 2022-11-23; First posted 2023-04-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Toric Intraocular Lens Stability; Visual Quality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cataract patients implanted with toric IOLs: Cataract patients who received the implantation of different toric IOLs with different haptic designs

SUMMARY:
This study included cataract patients who underwent toric intraocular lens (IOL) implantation, which aimed to evaluate the stability and clinical visual quality of toric IOLs.

DETAILED DESCRIPTION:
This study included cataract patients who underwent the implantation of toric intraocular lens (IOL) with haptic design, which aimed to evaluate the stability and clinical visual quality of toric IOLs.

ELIGIBILITY:
Inclusion Criteria:

* Cataract

Exclusion Criteria:

* • small pupil

  * zonular dehiscence
  * preexisting corneal pathology
  * glaucoma
  * uveitis
  * a history of ocular trauma or surgery
  * severe intraoperative and postoperative complications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cataract patients who underwent uneventful lens phacoemulsification and toric IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
IOL rotation degree at one hour | one hour
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at one day | one day
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at three days | three days
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at one week | one week
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at two weeks | two weeks
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at one month | one month
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at three months | three months
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at six months | six months
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at one year | one year
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL rotation degree at three years | three years
  After the pupil was dilated, the IOL axis was recorded using the same slit-lamp microscope. IOL rotation was defined as the difference between the target and final axis.
IOL tilt at one week | one week
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at two weeks | two weeks
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at one month | one month
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at three months | three months
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at six months | six months
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at one year | one year
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL tilt at three years | three years
  The tilt data were obtained from the wavefront mode of the OPD-Scan III aberrometer.
IOL decentration at one week | one week
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at two weeks | two weeks
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at one month | one month
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at three months | three months
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at six months | six months
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at one year | one year
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.
IOL decentration at three years | three years
  Decentration was defned as the distance between the center of the toric IOL and the visual axis and was calculated using Adobe Photoshop software on the retro image exported from the OPD-scan aberrometer.

SECONDARY OUTCOMES:
visual quality at one week | one week
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at two weeks | two weeks
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at one month | one month
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at three months | three months
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at six months | six months
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at one year | one year
  visual acuity was evaluated by OPD-Scan III aberrometer.
visual quality at three years | three years
  visual acuity was evaluated by OPD-Scan III aberrometer.

OTHER OUTCOMES:
visual acuity at one day | one day
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at one day
visual acuity at three days | three days
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at three days
visual acuity at one week | one week
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at one week
visual acuity at two weeks | two weeks
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at two weeks
visual acuity at one month | one month
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at one month
visual acuity at three months | three months
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at three months
visual acuity at six months | six months
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at six months
visual acuity at one year | one year
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at one year
visual acuity at three years | three years
  uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) were recorded after surgery at three years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, PhD, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (2):
- China (2):
  - Eye & ENT Hospital of Fudan University, Shanghai, China
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided